CLINICAL TRIAL: NCT05550506
Title: The Effect of Duloxetine on Bone Metabolism
Brief Title: Duloxetine on Bone Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Bayram Kelle, Associate Professor, Cukurova University
Other Study IDs: Duloxetine on Bone Metabolism
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain; Fibromyalgia
Keywords: duloxetine; chronic pain; fibromyalgia; bone metabolism
MeSH Terms: conditions — Chronic Pain; Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Duloxetine Group: Patients who use duloxetine at least 3 months for chronic pain or fibromyalgia
  Interventions: Drug: Duloxetine
- Healthy Group: Age and sex matched 51 healthy individuals

INTERVENTIONS:
Drug: Duloxetine — Patients who use duloxetine for chronic pain or fibromyalgia
  Groups: Duloxetine Group

SUMMARY:
The aim of the study was to determine the effect of duloxetine as monotherapy on biochemical markers and bone mineral density.

DETAILED DESCRIPTION:
51 patients diagnosed with chronic pain or fibromyalgia syndrome who were using duloxetine for at least 3 months and age and sex matched 51 healthy individuals were recruited for this cross-sectional study. Bone mineral density of both groups were measured by dual energy x ray absorbsiometry(DXA), bone biochemical markers, serum calcium, and vitamin D levels were investigated.

ELIGIBILITY:
Inclusion Criteria:

* >18 years or <50 years
* patients using duloxetine for at least 3 months due to chronic pain or fibromyalgia

Exclusion Criteria:

* postmenopausal women
* clinical conditions which cause secondary osteoporosis
* patients using medication that cause secondary osteoporosis
* pregnancy and malignity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who use duloxetine for at least 3 months due to chronic pain or fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
DXA | 3 months
  Bone mineral densitomtry
CTX | 3 months
  C-terminal telopeptide
OC | 3 months
  Osteocalcin
25-OH VITD3 | 3 months
  25-hydroxyvitamin D3

CONTACTS AND LOCATIONS:
Overall Officials: Burak Demir, Dr., Principal Investigator — Cukurova University Faculty of Medicine Department of Physical Medicine and Rehabilitation
Locations (1):
- Çukurova Üniversitesi, Adana, Turkey (Türkiye)